CLINICAL TRIAL: NCT07036965
Title: Comparison of Different Pulsed Field Ablation Catheters Combined With Stroke Prevention in High Stroke Risk·Atrial Fibrillation: A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Comparison of Different Pulsed Field Ablation Catheters in Atrial Fibrillation
Acronym: COMBINATION 2P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Dinova EP Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-IIS-007
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; pulsed field ablation; LAAC
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CardiPulse Group (Experimental): Patients accept atrial fibrillation ablation with CardiPulse pulsed field ablation catheter
  Interventions: Device: CardiPulse
- FaraPulse Group (Active Comparator): Patients accept atrial fibrillation ablation with FaraPulse pulsed field ablation catheter
  Interventions: Device: FaraPulse

INTERVENTIONS:
Device: CardiPulse — abc
  Arms: CardiPulse Group
Device: FaraPulse — bcd
  Arms: FaraPulse Group

SUMMARY:
Pulsed field energy ablation, a non-thermal ablation modality, can potentially reduce post-ablation tissue edema. Previous studies have confirmed the feasibility and safety of combined pulsed field ablation (PFA) and left atrial appendage closure (LAAC) as a one-stop treatment, with few reports of post-ablation tissue edema. However, during PFA procedures, the presence of metallic components in the ablation site (e.g., occluder frames, metallic valves) may lead to arcing during energy delivery, compromising procedural safety. Therefore, when performing PFA+LAAC as a one-stop procedure, a "ablation-first" strategy is recommended. Due to the influence of parameters such as voltage, pulse width, and number of cycles on pulsed field energy characteristics, significant variability in ablation depth and area may exist between different PFA devices. To date, no large-scale clinical studies have compared the efficacy and safety of different PFA systems. Accordingly, this study will conduct a prospective, multicenter, randomized controlled trial to compare the effectiveness and safety of domestic versus imported pulsed field ablation catheters in the treatment of patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years.
2. Diagnosed with drug-refractory, symptomatic atrial fibrillation.
3. The patient has a high risk of stroke (CHA2DS2-VA score ≥ 2).
4. Have a situation of:

   1. requires oral anticoagulation therapy
   2. high bleeding risk (HAS-BLED score ≥ 3) that unsuitable for or unwilling to undergo long-term oral anticoagulation therapy.
5. Subjects are able to understand the purpose of the study, voluntarily participate in the study and sign the informed consent, and are willing to complete the follow-up according to the requirements of the program.

Exclusion Criteria:

1. History of persistent atrial fibrillation >1 year.
2. Atrial fibrillation was secondary to thyroid disease or other reversible reasons.
3. Left atrial anteroposterior diameter >50 mm.
4. Evidence of left atrial or left atrial appendage thrombus on imaging examination.
5. Concurrent other arrhythmias required for catheter ablation (e.g., atrioventricular reentrant tachycardia, atrioventricular nodal reentrant tachycardia, pre-excitation syndrome) prior to enrollment.
6. Rheumatic heart disease.
7. Left ventricular ejection fraction <40% or New York Heart Association (NYHA) class III/IV.
8. Unstable angina.
9. Myocardial infarction (MI), coronary artery bypass grafting (CABG), or percutaneous coronary intervention (PCI) within 3 months prior to enrollment.
10. History of prior left atrial appendage closure, patent foramen ovale closure, atrial septal defect closure, or repair surgery.
11. Implantation of a mechanical mitral valve prosthesis or metallic annuloplasty rings.
12. Presence of intracardiac thrombus, space-occupying lesions, or other abnormalities that preclude vascular access or catheter manipulation.
13. Contraindications to anticoagulation or history of coagulation disorders/abnormal bleeding.
14. Active systemic infection.
15. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m² or history of renal dialysis.
16. Pregnancy or breastfeeding.
17. Life expectancy <12 months (e.g., advanced malignancy).
18. Current or anticipated participation in other drug or device clinical trials.
19. Any other condition or abnormality deemed by the investigator to warrant exclusion.

Min Age: 118 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
12-month atrial fibrillation (AF) ablation success rate | 12 months post-procedure
  Defined as the absence of AF, atrial flutter (AFL), or atrial tachycardia (AT) episodes ≥30 seconds on dynamic electrocardiogram (ECG) monitoring after the blanking period (90 days post-catheter ablation)

SECONDARY OUTCOMES:
Acute pulmonary vein ablation success rate | Immediately post-procedure
  Defined as maintained bidirectional block across the ablation line 20 minutes after ablation
Incidence of major adverse events (MAEs) related to the device | Within 7 days post-procedure
  Including stroke/transient ischemic attack (TIA), pulmonary vein stenosis, phrenic nerve paralysis, systemic embolism, pericarditis, pericardial effusion/cardiac tamponade, atrioesophageal fistula, myocardial infarction, or severe vascular access complications
Incidence of repeat ablation | Within 12 months post-procedure
  Summary ncidence of repeat ablation after the blanking period
AF burden | 6 and 12 months post-procedure
  Record AF burden at 6 and 12 months post-procedure
Incidence of cardiovascular MAEs | Within 12 months post-procedure
  Incidence of thromboembolic events (including stroke/TIA), cardiovascular-related rehospitalization, or cardiovascular mortality within 12 months post-procedure
Technical success rate of LAAC | Immediately post-procedure
  Defined as successful LAA occlusion without residual shunt >3 mm and no device-related complications
LAA closure rate | 3 and 6 months post-procedure
  Defined as imaging-confirmed residual shunt ≤3 mm at the device edges.
Incidence of new residual shunt | 3 and 6 months post-procedure
  Defined as any increase in residual shunt (post-procedure shunt volume - intraoperative shunt volume >0 mm)
Incidence of device-related thrombus | Within 12 months post-procedure.
  Record device-related thrombus events during follow-up
Discontinuation rate of anticoagulants and antiarrhythmic medications | Within 12 months post-procedure
  Record drugs history during follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo First Hospital, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No